CLINICAL TRIAL: NCT01008280
Title: Efficacy & Safety of Baclofen to Reduce Alcohol Use in Veterans With HCV
Brief Title: Baclofen to Reduce Alcohol Use in Veterans With HCV
Acronym: BRAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-014-09S
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C; Alcohol Use Disorders
MeSH Terms: conditions — Hepatitis C; Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Experimental): baclofen 10 mg po tid
  Interventions: Drug: baclofen
- Placebo (Placebo Comparator): placebo given tid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: baclofen — baclofen 10 mg tid
  Arms: Baclofen
Drug: placebo — placebo pill tid
  Arms: Placebo

SUMMARY:
Hepatitis C (HCV) is the most common blood born virus in the United States, affecting 1.8% of the general population and more than 5% of Veterans using VA facilities. As Veterans with HCV have high rates of co-morbid alcohol use disorders that accelerate greatly the liver damage caused by HCV, a safe and effective treatment for alcohol use disorders is needed. Baclofen is a novel treatment for alcohol use disorders that has minimal effect on the liver and may represent a safe and efficacious treatment option for Veterans with HCV and co-morbid alcohol use disorders.

DETAILED DESCRIPTION:
Project: Efficacy of baclofen in reducing alcohol consumption in Veterans with HCV Principal Investigator: Peter Hauser, MD

Keywords: Hepatitis C, Substance-Related Disorders, Alcoholism

Abstract

PLAN/METHODS: Two sites of the national VA Hepatitis C Resource Center, including Minneapolis and Portland VA Medical Centers (VAMCs), the Long Beach VAMC, and the San Diego VAMC (total 4 sites) will recruit 180 men, women, and minority Veterans who are HCV positive and currently drinking alcohol. Participants will be assessed for current alcohol use and alcohol use disorders and enrolled in the study if they meet eligibility criteria, mainly that they are drinking more than 7 drinks a week or have one heavy drinking day a week for the preceding two weeks. Enrolled subjects will be randomly assigned to one of two groups: Experimental group (Baclofen) or control (placebo). Subjects will be followed for a total of 14 weeks, and follow-up data will be collected at a total of 11 visits (weeks 1,2,3,4,6,8,10,12, and 14). At each visit, interviews will be conducted by a blinded interviewer assessing current stage of change and current alcohol use along with any changes in mood and psychological or somatic symptoms. HCV viral titers will be obtained at baseline and again at week 12 to determine the effect of abstinence on this measure. Data will also be collected from participants' medical records regarding enrollment and attendance in substance abuse treatment or self-help programs (Alcoholics Anonymous). Data will be analyzed using repeated measure ANOVAs to compare the groups on alcohol use and stage of change.

CLINICAL RELEVANCE: This study focuses on a current Veterans Health Administration (VHA) priority: treatment of Veterans with HCV. Alcohol use in this population is a major risk factor for progression of liver disease. The investigators anticipate that the Baclofen proposed in this study will result in reduced alcohol use, which is expected to result in a slowing of the progression of liver disease, improvement in physical health, and a reduction in long-term service utilization and mortality rates.

POTENTIAL IMPACT ON VETERANS HEALTH CARE: Effectively addressing alcohol use disorders in a hepatitis clinic will contribute to a new standard of care for HCV patients within the VA. Co-located care for patients with comorbid medical and substance use disorders is likely to improve access to effective treatment, acceptance by patients and improve clinical efficiency.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Participation Include if:

* Male or female
* Age 18 or older

Medical record shows:

* Serum antibody positive for HCV and PCR (Polymerase Chain Reaction) confirmation, Men or Women: > 7 drinks per week for each of the proceeding 2 weeks Or One heavy drinking day per week for 2 weeks (Heavy drinking day: 5 drinks in one day for men and >4 drinks in one day for women) based on Timeline Followback method (TLFB)
* Alcohol use Disorder (abuse or dependence) based on Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID)

  * Yes Medical record and self report
  * Medical record, self report, SCID, Beck Depression Inventory -II (BDI-II)
  * Able to attend clinic appointments
  * Yes No Self-report

Exclusion Criteria:

Criteria for Participation Exclude if:

* Male or female
* Under age 18
* Cocaine, methamphetamine or opioid dependence within the past 6 months*
* Any known pre-existing medical conditions that could interfere with participation in the protocol, such as:

  * Central Nervous System (CNS) trauma
  * Known cognitive impairment
  * Dementia
  * Encephalopathy from liver disease
  * Acute psychiatric instability, such as significant psychosis, mania, or elevated risk for suicide
* Not able to attend clinic appointments
* Pregnant women
* If any of the following medication are being used:

  * Ondansetron
  * Disulfiram
  * Topiramate
  * Naltrexone
  * Acamprosate
  * Buprenorphine
  * Methadone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hauser, MD, Principal Investigator — VA Long Beach Healthcare System, Long Beach, CA
Locations (4):
- United States (4):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Portland, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baclofen | Placebo
Started | 88 | 92
Completed | 67 | 73
Not Completed | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen | Placebo | Total
Number analyzed (Participants) | 88 | 92 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (7.1) | 57.5 (6.9) | 56.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 85 | 92 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 70 | 76 | 146
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 31 | 35 | 66
  White | 52 | 50 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days in the Past Two Weeks
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: Number of Drinking Days/2 weeks
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 88 | 92
Number of Drinking Days/2 weeks
  Baseline | 8.6 (.50) | 8.9 (.45)
  Weeks 0-1 | 6.8 (.55) | 7.1 (.54)
  Weeks 2-3 | 6.2 (.55) | 6.3 (.55)
  Weeks 4-5 | 5.7 (.57) | 5.8 (.58)
  Weeks 6-7 | 5.4 (.57) | 5.4 (.59)
  Weeks 8-9 | 5.1 (.58) | 4.8 (.59)
  Weeks 10-11 | 4.6 (.55) | 4.7 (.63)
Statistical Analysis 1: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed time effects for the number of drinking days; Test type: Superiority or Other; p < 0.01, Wald Chi-squared
Statistical Analysis 2: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed group effects for the number of drinking days; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared
Statistical Analysis 3: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed time by group effects for the number of drinking days; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared

2. Primary Outcome: Number of Drinks Consumed Per Two Week Segments
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Number of Drinks/2 Weeks
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 88 | 92
Number of Drinks/2 Weeks
  Baseline | 60.09 (5.04) | 67.23 (5.09)
  Weeks 0-1 | 41.89 (4.42) | 47.68 (4.97)
  Weeks 2-3 | 33.88 (4.32) | 39.07 (4.52)
  Weeks 4-5 | 28.46 (3.62) | 37.73 (5.65)
  Weeks 6-7 | 31.82 (5.54) | 30.73 (5.04)
  Weeks 8-9 | 26.01 (4.59) | 26.69 (4.36)
  Weeks 10-11 | 18.82 (2.67) | 22.85 (3.71)
Statistical Analysis 1: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed time effects for the number of drinks; Test type: Superiority or Other; p < 0.01, Wald Chi-Squared
Statistical Analysis 2: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed group effects for the number of drinks; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared
Statistical Analysis 3: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed group by time effects for the number of drinks; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared

3. Primary Outcome: Number of Heavy Drinking Days Per Two Week Segment
Description: A heavy drinking day was defined as ≥4 drinks/ day if female or ≥5 drinks/day if male
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Number of heavy drinking days/2 weeks
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 88 | 92
Number of heavy drinking days/2 weeks
  Baseline | 6.48 (.53) | 7.18 (.51)
  Weeks 0-1 | 3.67 (.46) | 4.04 (.46)
  Weeks 2-3 | 2.59 (.37) | 3.07 (.41)
  Weeks 4-5 | 2.40 (.38) | 3.29 (.50)
  Weeks 6-7 | 2.52 (.46) | 2.44 (.44)
  Weeks 8-9 | 2.10 (.46) | 2.18 (.42)
  Weeks 10-11 | 1.37 (.31) | 2.15 (.46)
Statistical Analysis 1: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed time effects for the number of heavy drinking days; Test type: Superiority or Other; p < 0.01, Wald Chi-Squared
Statistical Analysis 2: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed group effects for the number of heavy drinking days; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared
Statistical Analysis 3: Comparison: Baclofen vs Placebo; This was an intent to treat analysis where Generalized Estimating Equations, using the Negative Binomial function, were used to test for group, time, and group by time effects for drinks, drinking days, and heavy drinking days. This analysis assessed group by time effects for the number of heavy drinking days; Test type: Superiority or Other; p > 0.01, Wald Chi-Squared

ADVERSE EVENTS:
Arm/Group | Baclofen | Placebo
Serious Adverse Events (participants affected / at risk) | 6/88 | 3/92
Other Adverse Events (participants affected / at risk) | 70/88 | 68/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen (N=88) | Placebo (N=92)
Dizziness, Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Subject stopped taking study medication and was discontinued from the study.
Mental Status Change (Psychiatric disorders) | 0 (0) | 1 (1) — Subject had an increase in BDI-II (Beck Depression Inventory-II) depression scores and mental status change.
Tightness in the head and Chest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject was hospitalized over night. Chest and head tightness was determined to be related to an epidural the patient received the day before.
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject was admitted for GI bleeding, needed 8 bands in the esophagus.
Substance Abuse/Intoxication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject was hospitalized after suspected mix of alcohol and opiate drugs.
Altered Mental Status and Renal Failure (Psychiatric disorders) | 1 (1) | 0 (0) — Subject was hospitalized two times, once for altered mental status and acute renal insufficiency, then again for alcohol withdrawal, hypertension and acute renal failure.
Alcohol Withdrawal Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject was hospitalized for Alcohol Withdrawal
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — subject was hospitalized for hypotension
Mild Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Subject had a preexisting history of chest pressure prior to participation in this study. Subject was withdrawn from the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baclofen (N=88) | Placebo (N=92)
Abdominal Pain (General disorders) | 12 | 15
Bedwetting (Renal and urinary disorders) | 5 | 1
Blurred Vision (Eye disorders) | 9 | 9
Confusion (General disorders) | 20 | 14
Constipation (General disorders) | 14 | 14
Depression (Psychiatric disorders) | 5 | 14
Diarrhea (Gastrointestinal disorders) | 8 | 20
Difficulty Breathing at Night (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Difficulty Moving (General disorders) | 10 | 6
Dizziness (General disorders) | 23 | 21
Double Vision (Eye disorders) | 4 | 3
Drowsiness (General disorders) | 34 | 30
Dry Mouth (General disorders) | 14 | 16
Excessive Perspiration (General disorders) | 13 | 10
Erectile Dysfunction (Reproductive system and breast disorders) | 5 | 7
Excitement (General disorders) | 9 | 11
Fatigue (General disorders) | 10 | 13
Hallucinations (Psychiatric disorders) | 5 | 3
Headache (General disorders) | 22 | 18
Heart Palpitations (Cardiac disorders) | 7 | 6
Hypotension (General disorders) | 7 | 0
Insomnia (Psychiatric disorders) | 8 | 18
Itching (General disorders) | 13 | 9
Lack of Coordination (General disorders) | 7 | 11
Loss of Appetite (General disorders) | 12 | 17
Loss of Consciousness (General disorders) | 4 | 2
Involuntary Muscle Movement (Musculoskeletal and connective tissue disorders) | 12 | 9
Muscle Pain (Musculoskeletal and connective tissue disorders) | 11 | 16
Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 14 | 11
Nasal Congestion (General disorders) | 11 | 13
Nausea (General disorders) | 14 | 22
Paresthesia (General disorders) | 11 | 1
Problems Speaking (General disorders) | 8 | 9
Rash (Skin and subcutaneous tissue disorders) | 8 | 3
Ringing in Ears (Ear and labyrinth disorders) | 4 | 8
Slurred Speech (General disorders) | 9 | 4
Swelling in Ankles (General disorders) | 4 | 2
Taste Disturbance (General disorders) | 5 | 5
Tremor (General disorders) | 6 | 7
Urinary Frequency (Renal and urinary disorders) | 11 | 15
Urinary Retention (Renal and urinary disorders) | 4 | 5
Vomiting (General disorders) | 8 | 11
Weakness (General disorders) | 13 | 15
Weight Gain (General disorders) | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No